CLINICAL TRIAL: NCT03747042
Title: Pre-Surgical Trial of Letrozole in Post-Menopausal Patients with Operable Hormone-Sensitive Breast Cancer
Brief Title: Letrozole in Post-Menopausal Patients with Operable Hormone-Sensitive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Nisha Unni, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCC-11118; STU-2018-0015
Record Dates: First submitted 2018-11-15; First posted 2018-11-20 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Female
Keywords: ER-positive; HER2-negative; invasive mammary carcinoma
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Drug: letrozole Take by mouth at a dose of 2.5 mg on days 7-30
  Other: Blood Collection Blood used for gene expression analysis and reverse transcriptase-polymerase chain reaction
  Procedure: biopsy/lumpectomy/mastectomy Tissue collection,Surgery to remove tumor, Tumor tissues used for laboratory biomarker analysis
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Patients will receive a prescription for letrozole to be taken orally for 7-30 days to allow for variations in surgical scheduling. Patients are to undergo surgical resection of their tumor the day after the last dose of letrozole. Post-treatment tumor biopsies (a goal of 4-6 cores) will be obtained following 7-56 days of letrozole treatment on the day of surgery.

SUMMARY:
A short pre-surgical non-therapeutic trial involving postmenopausal women with newly diagnosed eR+, HeR2-negative operable breast cancers. After undergoing a core needle biopsy for tissue acquisition, study participants will take a 7- to 30-day (1-4 weeks) course of letrozole in accordance with standard of care. They will then undergo definitive surgical resection of their primary tumor (mastectomy vs lumpectomy) as per standard of care guidelines.

DETAILED DESCRIPTION:
Patients will receive a prescription for letrozole to be taken orally at a dose of 2.5 mg/day for 7-30 days to allow for variations in surgical scheduling. Patients are to undergo surgical resection of their tumor the day after the last dose of letrozole.

Post-treatment tumor biopsies (a goal of 4-6 cores) will be obtained following 7-30 days of letrozole treatment on the day of surgery. Frozen AND formalin fixed core biopsies will be obtained whenever possible. The tissue will be used for study-specific assays as well as routine histopathology. Post-treatment core needle biopsy tissue will be obtained, whenever possible, by the surgeon intraoperatively at the time of routine surgical resection. A formalin-fixed paraffin embedded tumor block from the patient's surgical resection is also requested. This block will be used for a subset of the correlative studies if no tumor is obtained by the post treatment core biopsies. This block will be returned to pathology promptly after the correlative studies are completed.

Surgical treatment (total mastectomy or segmental resection with lymph node evaluation if clinically indicated) will occur the day after completion of therapy.

The primary lesion obtained at the time of the definitive surgical procedure (partial or total mastectomy) will be sent for standard of care histopathologic analysis; wherever possible intra-opearative cores from the central portion of the tumor will be obtained for study-specific assays. All specimens will be handled according to established institutional guidelines to maintain the accuracy of the analysis of tumor size and margin status.

Following standard of care histopathologic analysis, additional paraffin-embedded sections will be submitted at a later time to the Simmons Cancer Tissue Core to determine tumor proliferation with Ki67 (MIB1Ab, Dako Cytomation) IHC. These tests are of no clinical utility and will be done for research purposes only.

Frozen cores and/or peels from the formalin-fixed paraffin-embedded (FFPE) tumor blocks from the surgical specimen will be selected and/or macrodissected - when needed - based on ≥20% tumor cellularity as assessed by Dr. Sahoo, expert breast pathologist in the trial. These will be sent to Dr. Carlos Arteaga's laboratory for further testing.

ELIGIBILITY:
Inclusion Criteria:

1. Eligibility waivers are not permitted. Subjects must meet all of the inclusion and exclusion criteria to be registered to the study. Study treatment may not begin until a subject is registered.
2. Patients must provide informed written consent
3. ECOG performance status 0-2.
4. Clinical stage operable I, II or III invasive mammary carcinoma, which is ER-positive by IHC and HER2-negative by Herceptest (0 or 1+) or not amplified by in situ hybridization as per routine clinical testing.

   * Patients who have measurable residual tumor at the primary site
   * Patients who will undergo surgical treatment with either segmental resection or total mastectomy
5. Measurable tumor. Measurable disease: a mass that can be reproducibly measured by physical exam, mammogram or ultrasound and is at least 1 cm in size
6. Post-menopausal female subjects ≥18 years of age, as defined by any of the following:

   * Subjects at least 55 years of age;
   * Subjects under 55 years of age and amenorrhoeic for at least 12 months or follicle-stimulating hormone (FSH) values ≥40 IU/L and estradiol levels ≤40 pg/mL (140 pmol/L) or in postmenopausal ranges per local or institutional reference ranges;
   * Prior bilateral oophorectomy or prior radiation castration with amenorrhea for at least 6 months.
   * (There is no upper age limit for enrollment to this study)
7. No prior chemotherapy for this primary breast cancer.
8. Patients with a prior history of contralateral breast cancer are eligible if they have no evidence of recurrence of their initial primary breast cancer.
9. Women may have been taking tamoxifen or raloxifene as a preventive agent prior to study entry but must have discontinued the drug for at least 14 days prior to study enrollment.
10. Subjects must have ended hormone replacement therapy (HRT) (e.g., conjugated estrogens tablets, USP, [Premarin]), at least 7 days prior to receiving the first dose of randomized therapy.
11. Patients must have adequate hepatic and renal function. All tests must be obtained less than 4 weeks from study entry. This includes:

    1. Creatinine <2X upper limits of normal
    2. Bilirubin, SGOT, SGPT <1.5X upper limits of normal
12. Able to swallow and retain oral medication

Exclusion Criteria:

1. Patients with locally advanced disease who are candidates for other preoperative chemotherapy at the time of initial evaluation. This may include patients with locally advanced disease such as:

   * Inflammatory breast cancer (T4d)
   * Fixed axillary lymph node metastases (N2)
   * Metastasis to ipsilateral internal mammary node (N3)
2. Locally recurrent breast cancer
3. Evidence of distant metastatic disease (i.e. lung, liver, bone, brain, etc.)
4. Serious medical illness that in the judgment of the treating physician places the patient at high risk of operative mortality.
5. Severe uncontrolled malabsorption condition or disease (i.e. grade II/III diarrhea, severe malnutrition, short gut syndrome)
6. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
7. Use of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of letrozole.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Measure Ki67 index in highly hormone-dependent breast cancers vs. those that are not | Within 8 to 30 days
  Ki67 index measured 1-4 weeks after therapy with letrozole to segregate hormone receptor-positive breast cancers that are highly hormone-dependent vs. those that are not

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Unni, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No